CLINICAL TRIAL: NCT03590886
Title: A Clinical Study About Gut Microbes and Metabolic Group in Different PBC Patients for UDCA Response
Brief Title: Gut Microbes and Metabolic Group in Different PBC Patients for UDCA Response
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, professor, Sun Yat-sen University
Other Study IDs: UDCA20181123
Record Dates: First submitted 2018-06-27; First posted 2018-07-18 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Primary Biliary Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- total response Group: The PBC patients show biochemical response for UDCA treatment more than 1 year according to Paris-I/II standard
  Interventions: Other: total response Group
- poor response group: The PBC patients show poor biochemical response for UDCA treatment more than 1 year according to Paris-I/II standard

INTERVENTIONS:
Other: total response Group — biochemical response for UDCA treatment more than 1 year according to Paris-I/II standard
  Other Names: poor response group
  Groups: total response Group

SUMMARY:
To compare intestinal flora diversity in different PBC patients with UDCA responses, and further study the differences of bile acid metabolism and short chain fatty acid metabolism in feces and serum of two groups of PBC patients.

DETAILED DESCRIPTION:
The PBC patients have been enrolled in the study for UDCA treatment more than 1 year, who is divided into the UDCA total response Group and the other poor response group according to Paris-I/II standard .The feces of two groups of patients were collected and the differences of microbial polymorphism of fecal microorganism in two groups were observed. The metabolic differences of bile acids and short chain fatty acids in serum and feces of two groups of PBC patients were studied by means of metabolic proteomics.

ELIGIBILITY:
Inclusion Criteria:

1.Confirmed diagnostic criteria about PBC, and orally UDCA treatment for more than a year; 2.30-70 years old; 3.Currently only UDCA therapy, not glucocorticoids and immunosuppressor treatment.

Exclusion Criteria:

1. Viral liver disease;
2. alcoholic liver disease;
3. fatty liver;
4. drug-associated liver damage;
5. infectious disease;
6. obesity;
7. gastrointestinal diseases;
8. combined with other autoimmune diseases;
9. cardiac and pulmonary dysfunction;
10. renal dysfunction, malignant tumor,;
11. neurological and psychiatric abnormalities;
12. nearly 2 months to take antibiotics and probiotics;
13. nearly 3 months participate in other drug clinical trials .

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary biliary cholangitis patients
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
fecal microbial diversity | 6 months
  Macrogenomic examination of fecal microbial DNA

SECONDARY OUTCOMES:
bile acid metabolites | 6 months
  The examination of bile acid metabolites by ELISA methods
short chain fatty acid metabolites | 6 months
  The examination of short chain fatty metabolites by ELISA methods

CONTACTS AND LOCATIONS:
Overall Officials: Lin B Liang, MD, Study Director — Third Affliated Hospital of Sun Yat-sen University
Locations (1):
- The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No